CLINICAL TRIAL: NCT01437449
Title: Weekly Docetaxel, Cisplatin, and Cetuximab (TPC) in Palliative Treatment of Patients With SCCHN
Brief Title: Docetaxel, Cisplatin, and Cetuximab (TPC) in Palliative Treatment of Patients With Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, A. Dimitrios Colevas, Professor of Medicine (Oncology) and Otolaryngology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-22329; SU-08222011-8290 (Other: Stanford University Medical Center); NCI-2011-03271 (Other: CTRP); ENT0033 (Other: OnCore)
Record Dates: First submitted 2011-09-16; First posted 2011-09-20 (Estimated); Results first posted 2019-12-17 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Head and Neck Cancer
Keywords: Quality of Life
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Docetaxel; Cisplatin; Cetuximab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cisplatin + Docetaxel + Cetuximab (Experimental): Patients will be treated weekly with cisplatin, docetaxel, and cetuximab.
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Drug: Cetuximab; Drug: Carboplatin

INTERVENTIONS:
Drug: Docetaxel — 30 mg/m² by intravenous (IV) administration
  Other Names: Taxotere
Drug: Cisplatin — 30 mg/m² by intravenous (IV) administration
  Other Names: Cisplatinum; Platinol
Drug: Cetuximab — 400 mg/m² by intravenous (IV) administration, thereafter 250 IV
  Other Names: Erbitux
Drug: Carboplatin — Area under the free carboplatin plasma concentration versus time curve (AUC)=2 by intravenous (IV) administration
  Other Names: Paraplatin

SUMMARY:
Docetaxel and cetuximab are FDA-approved for the treatment of squamous cell carcinoma of the head and neck (SCCHN). Cisplatin and carboplatin, while not FDA-approved for SCCHN, have been used as standard of care in SCCHN patients in combination with other drugs. This study evaluates if weekly cisplatin and docetaxel, in combination with cetuximab, is effective in palliative treatment of patients with SCCHN. These drugs will be given intravenously weekly, repeated 3 of every 4 weeks until evidence of disease progression or unacceptable adverse events.

DETAILED DESCRIPTION:
Primary Objective:To establish the response rate using RECIST 1 criteria to weekly TPC in patients with metastatic or relapsed squamous cell carcinoma of the head and neck Secondary Objective: To establish the safety profile, progression free and overall survival of weekly TPC in this patient population.

ELIGIBILITY:
INCLUSION CRITERIA

* Squamous cell carcinoma (SCC) of head and neck (SCCHN), including all pharynx, larynx, oral cavity, skin and para-nasal sinus sites. Patients with SCC of unknown primary presenting in the neck clinically compatible with head and neck mucosal primary sites are eligible.
* If prior chemoradiation, radiation, and/or surgery in the potentially curative setting, > 3 months has elapsed since the end of the potentially curative treatment ended
* If history of other malignancies treated curatively > 1 year prior to enrollment, no evidence of relapse at the time of enrollment
* If brain metastasis, central nervous system (CNS) imaging documents no evidence of CNS progression at least 30 days following definitive CNS treatment (resection or radiation)
* ≥ 16 years old
* Eastern cooperative oncology group (ECOG) Performance Status < 3
* Laboratory value requirements at enrollment:
* Absolute neutrophil count > 1500/mm³
* Platelet count > 100,000/mm³
* Hemoglobin > 8 g/dL
* Aspartate aminotransferase (AST) / alanine aminotransferase (ALT) < 2.5 x upper limit of normal (ULN) unless liver metastases documented. If so, AST and ALT < 5 x ULN required.
* Total bilirubin < 1.5 x ULN, EXCEPT if Gilbert's syndrome is present. If so, total bilirubin < 2.5 x ULN
* Serum Creatinine < 1.5 mg/dL OR an estimated creatinine clearance from 24 hour urine collection > 50 mL/min
* Peripheral neuropathy < grade 2
* Hearing loss in best ear < grade 2 per Chang criteria if audiogram performed. Formal audiology is not required in patients with no clinical evidence of hearing loss at baseline.
* Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA

* Prior palliative chemotherapy
* Active infections including HIV (EXCEPTION: HIV-positive patients on HAART with undetectable blood HIV levels, or with history or serological evidence of exposure to Hepatitis B without active infection are eligible)
* Prior grade 3 allergic or infusion reactions to docetaxel, cisplatin or cetuximab (EXCEPTION: a history of infusion reactions that were well-tolerated, at physician's discretion)
* Pregnant and/or lactating

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-10; Primary Completion 2018-09-11 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. Dimitrios Colevas, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - University of California Davis Medical Center, Davis, California
  - Stanford University, School of Medicine, Stanford, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Trieu V, Pinto H, Riess JW, Lira R, Luciano R, Coty J, Boothroyd D, Colevas AD. Weekly Docetaxel, Cisplatin, and Cetuximab in Palliative Treatment of Patients with Squamous Cell Carcinoma of the Head and Neck. Oncologist. 2018 Jul;23(7):764-e86. doi: 10.1634/theoncologist.2017-0618. Epub 2018 Mar 14. PMID 29540603

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cisplatin + Docetaxel + Cetuximab
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cisplatin + Docetaxel + Cetuximab
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Clinical response for each participant will be assessed after 8 weeks of treatment according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria. Overall response rate (ORR) was assessed as the sum of the number of participants that experience a complete response (CR) or partial response (PR). The outcome is defined and reported as the number of subjects that responded, a number without dispersion. Other response statuses are included. RECIST v1.1 criteria is defined as follows.
  * Complete Response (CR) = Disappearance of all target lesions
  * Partial Response (PR) = ≥ 30% decrease in the sum of the longest diameter of target lesions
  * Overall Response (OR) = CR + PR
  * Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions, and/or the appearance of one or more new lesion(s)
  * Stable disease (SD) = Small changes that do not meet any of the above criteria
Time Frame: 8 weeks
Population: Response data were not available for all participants.
Measure: Number; unit: participants
Arm/Group | Cisplatin + Docetaxel + Cetuximab
Number analyzed (Participants) | 26
participants
  Complete Response (CR) | 1
  Partial Response (PR) | 14
  Overall Response (OR) | 15
  Stable disease (SD) | 5
  Progressive disease (PD) | 6

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS), defined as the duration of time from start of treatment to time of progression or death, was assessed through 24 months, according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria. The outcome is reported as the median time that participants remained free of progression, with 95% confidence interval (CI).
  * Complete Response (CR) = Disappearance of all target lesions
  * Partial Response (PR) = ≥ 30% decrease in the sum of the longest diameter of target lesions
  * Overall Response (OR) = CR + PR
  * Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions, and/or the appearance of one or more new lesion(s)
  * Stable disease (SD) = Small changes that do not meet any of the above criteria
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cisplatin + Docetaxel + Cetuximab
Number analyzed (Participants) | 27
months | 4.8 [2.7 to 6.6]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was assessed through 24 months. The outcome is reported as the median time that participants remained alive, with 95% CI.
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cisplatin + Docetaxel + Cetuximab
Number analyzed (Participants) | 27
months | 14.7 [8.3 to NA] — The upper limit of the 95% confidence interval has not been reached.

4. Secondary Outcome: Grade 3, 4, and 5 Related Adverse Events (Toxicities)
Description: Related adverse events are considered toxicities. The outcome was assessed as adverse events and serious adverse events (SAEs per 21CFR§312.32) at least Grade 3, and are reported as the number of toxicities by grade (3, 4 or 5), a number without dispersion.
Time Frame: 2 years
Measure: Number; unit: Related Adverse Events
Arm/Group | Cisplatin + Docetaxel + Cetuximab
Number analyzed (Participants) | 27
Related Adverse Events | 24

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Cisplatin + Docetaxel + Cetuximab
All-Cause Mortality (participants affected / at risk) | 13/27
Serious Adverse Events (participants affected / at risk) | 27/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cisplatin + Docetaxel + Cetuximab (N=27)
Colitis (Gastrointestinal disorders) | 1 (4)
Gastrointestinal disorders - Other, Oral cavity infection (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, Pneumoperitoneum,Pneumoperitoneum (Gastrointestinal disorders) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 2 (3)
Facial pain (General disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, Abdominal wall infection associated with G-Tube- Recovering (Infections and infestations) | 1 (2)
Sepsis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Failure to thrive (Musculoskeletal and connective tissue disorders) | 2 (3)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Nervous system disorders - Other, Neurological deficit (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (3)
Bladder perforation (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other,Penile pain (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, Complicated urinary tract infection (UTI) (Renal and urinary disorders) | 1 (1)
Aspiration/Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory, thoracic and mediastinal disorders - Other, Air obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, CAP (pneumonia) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Right hand abscess (Skin and subcutaneous tissue disorders) | 1 (1)
Surgical and medical procedures - Other, G-Tube fell out & replacement (Surgical and medical procedures) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
Neoplasms benign, malignant. and unspecified (incl cysts and polyps) - Other, disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cisplatin + Docetaxel + Cetuximab (N=27)
Lymphocyte count decreased (Investigations) | 19 (104)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Abdominal infection (Infections and infestations) | 1 (1)
White blood cell decreased (Investigations) | 4 (5)
Syncope (Nervous system disorders) | 1 (2)
Alkaline phosphatase increase (Investigations) | 1 (1)
Aspartate aminotransferase increase (Investigations) | 1 (1)
Alanine aminotransferase increase (Investigations) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (16)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorders -Other, mouth sores (Gastrointestinal disorders) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (4)
Blurred vision (Eye disorders) | 1 (1)
Fatigue (General disorders) | 4 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Dizziness (Nervous system disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (3)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (3)
Neuropathy (Nervous system disorders) | 1 (1)
INR increased (Investigations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Hypocalcemia (Investigations) | 1 (2)
Catheter related infection (Infections and infestations) | 1 (2)
Pain (General disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Acute Kidney injury (Renal and urinary disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Respiratory, thoracic and mediastinal disorders, others, hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
General disorders and administration site conditions, others- failure to thrive (General disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-26): https://cdn.clinicaltrials.gov/large-docs/49/NCT01437449/Prot_SAP_000.pdf